CLINICAL TRIAL: NCT03354806
Title: Peripheral Analgesia in Painful Diabetic Neuropathy
Acronym: DIALOXY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: january 2019
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/CHU/05
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Neuropathy Peripheral; Neuropathic Pain; Diabetic Foot Infection
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Comparative, monocentric study including 2 parallel groups. Patient's allocation is based on recommended criteria for catheters for continuous peripheral nerve blocks uses such as anlagesic treatment (ropivacain) tolerance and acceptance or analgesic treatment refusal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous peripheral nerve blocks (Experimental): Ropivacaine-continous treatment using catheters for continous sciatic nerve blocks
  Interventions: Procedure: Continuous peripheral nerve blocks
- Analgesic treatment (Active Comparator): Pharmacological pain management in accordance with WHO's pain relief ladder
  Interventions: Procedure: Analgesic treatment

INTERVENTIONS:
Procedure: Continuous peripheral nerve blocks — 6 weeks-ropivacaine treatment delivered by continuous peripheral nerve blocks Transcutaneous oxygen measurement is assessed on day 2, week 3 and week 6 under atmospheric and hyperbaric conditions
  Arms: Continuous peripheral nerve blocks
Procedure: Analgesic treatment — 6 weeks-analgesic treatment according to WHO's pain relief ladder Transcutaneous oxygen measurement is assessed on day 2, week 3 and week 6 under atmospheric and hyperbaric conditions
  Arms: Analgesic treatment

SUMMARY:
Chronic obliterative arteriopathy of the inferior limbs is a frequent condition observed in diabetics. The later stages induce pain at rest and trophic disorders (ulcer, gangrene) that lead to chronic limb ischemia. Without possible surgical revascularization ,pain management and tissue healing are used to avoid amputation.

Prevalence of diabetes is twice higher in Reunion Island than in metropolitan France. As a consequence, the rate co-morbobidities, such as chronic obliterative arteriopathy of the inferior limbs, is also increases.

This study compares the efficiency of two analgesic treatments in diabetics with forefoot injuries.

DETAILED DESCRIPTION:
Patients are allocated in two groups regarding :

* their eligibility to analgesic treatment using continuous peripheral nerve blocks
* the unability of usual pain management to reduce their pain (pain visual analogic scale equal to or more than 4).

When patient 's response to pharmacological analgesic treatment is sufficient (pain visual analogic scale equal to or less than 3), patient is allocated to the control group.

Patients of experimental group received a continous analgesic treatment for 6 weeks using ropivacaine (2mg/ml, flow rate 7 ml/h).

Patients of control group received an analgesic treatment according the recommended pain ladder of World Health Organization (WHO). Opioids for mild-to-moderate pain are used in combination with a non-opioid analgesic, such as paracetamol, at the second step of the ladder. If regular maximum doses of opioids for mild-to-moderate pain do not achieve adequate analgesia, then they should be replaced with an opioid for moderate-to-severe pain, such as morphine.

Efficiency of both treatment is assessed the improvement of oxygen level in the tissue below the skin of the injured forefoot through the study.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient
* Diabetics with chronic obliterative arteriopathy of the inferior limbs
* Permanent limb ischaemia with a TcPO2 of the front-foot of at least 10 mmHg under atmospheric conditions
* Lack of surgical revascularization
* No contraindication to hyperbaric therapy
* Signed informed consent

Exclusion Criteria:

* Contraindication to ropivacaine
* Conditions that could alter hyperbaric measurements (anemia < 8 g/dl, cardiac or respiratory insufficiency)
* patients with planned limb amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Foot tissue oxygenation on day 2 | on day 2
  Measurement of transcutaneous oxygen tension (TcPO2) at room conditions

SECONDARY OUTCOMES:
Foot tissue oxygenation in hyperaemia-induced condition on day 2 | on day 2
  Measurement of transcutaneous oxygen tension (TcPO2) under hyperbaric conditions
Foot tissue oxygenation on week 6 | on week 6
  Measurement of transcutaneous oxygen tension (TcPO2) at room conditions
Foot tissue oxygenation in hyperaemia-induced condition on day 2 | on week 6
  Measurement of transcutaneous oxygen tension (TcPO2) under hyperbaric conditions

CONTACTS AND LOCATIONS:
Overall Officials: Valérie NAKAMURA, MD, Principal Investigator — Centre Hpospitalier Universitaire de La REUNION